CLINICAL TRIAL: NCT02045485
Title: Increased Risk of Atrial and Ventricular Arrhythmia in Long-lasting Psoriasis
Brief Title: P Wave and QT Dispersion in Psoriasis
Status: Completed | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, hakki simsek, Assistant proffessor, Yuzuncu Yil University
Other Study IDs: 901215
Record Dates: First submitted 2013-02-26; First posted 2014-01-24 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Arrhytmia in Psoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Background:

Several reports have demonstrated an association between psoriasis and cardiovascular diseases. P wave dispersion (PWD) is the most important electrocardiographic (ECG) markers used to evaluate the risk of atrial arrhythmias. QT dispersion (QTD) can be used to assess homogeneity of cardiac repolarization and may be a risk for ventricular arrhythmias.

Aim: To search PWD and QTD in patients with psoriasis. Methods: Ninety-four outpatient psoriasis patients and 51 healthy people were evaluated by physical examination, 12-lead ECG and transthoracic echocardiography. Severity of the psoriasis was evaluated by psoriasis Area and Severity Index (PASI).

DETAILED DESCRIPTION:
Ninety-four outpatient psoriasis patients and 51 healthy people were included in the study. Patients having systemic hypertension, diabetes mellitus, history of ischemic heart disease, significant valvular heart disease, chronic obstructive pulmonary disease, hypo or hyper-thyroidism, renal failure or any associated systemic disease were excluded. Diagnosis of psoriasis was confirmed by dermatological examination and/or punch biopsy. Severity of the psoriasis was evaluated by psoriasis area and severity index (PASI). Patients were evaluated by physical examination, 12-lead electrocardiography and transthoracic echocardiography.

ELIGIBILITY:
Patients having systemic hypertension, diabetes mellitus, history of ischemic heart disease, significant valvular heart disease, chronic obstructive pulmonary disease, hypo or hyper-thyroidism, renal failure or any associated systemic disease were excluded.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diagnosis of psoriasis was confirmed by dermatological examination and/or punch biopsy.
Sampling Method: Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2006-01; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
duration of p wave and QT interval | 3 -360 months